CLINICAL TRIAL: NCT01668524
Title: A Phase 2a Open-Label, Dose-ranging Study of the Safety and Tolerability of ATS907 in Subjects With Primary Open Angle Glaucoma and Ocular Hypertension
Brief Title: ATS907 Ph2a Open-Label Dose-ranging Safety and Tolerability in Primary Open Angle Glaucoma (POAG) and Ocular Hypertension (OHT) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altheos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATS907-205
Record Dates: First submitted 2012-08-14; First posted 2012-08-20 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm: ATS907 (Experimental): Single-cohort, dose-escalation
  Interventions: Drug: ATS907

INTERVENTIONS:
Drug: ATS907 — Single dose of each of three increasing concentrations

SUMMARY:
This single-site, dose-escalation study will evaluate safety and tolerability of increasing concentrations of ATS907 in 12 subjects with Primary Open Angle Glaucoma and/or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Diagnosis of open angle glaucoma or ocular hypertension in both eyes
* Corrected visual acuity in each eye +1.0 logMAR or better by Early Treatment Diabetic Retinopathy Study (EDTRS) in each eye (equivalent to 20/200)
* Must be willing to discontinue the use of all ocular hypotensive medications in both eyes prior to and during the entire course of the study

Exclusion Criteria:

Ophthalmic (in either eye):

* Glaucoma: pseudoexfoliation, steroid induced, pigment dispersion glaucoma, and or history of angle closure. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s). Refractive surgery in study eye
* Cataract surgery and or other intraocular surgery within one month prior to Screening in either eye
* History within 3 months prior to Screening of clinically significant moderate or severe chronic or active ocular infection, inflammation, blepharitis, dermatitis, uveitis or conjunctivitis
* Clinically significant corneal dystrophy, epithelial and or endothelial disease, corneal irregularities and or scarring such that reliable applanation tonometry would prevented
* Contact lens wear during the duration of the study
* Clinically significant ocular disease (e.g., diabetic retinopathy, macular degeneration, or uveitis) which might interfere or progress during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Evaluate local ocular safety and tolerability: change from baseline in ocular tolerability signs and symptoms (hyperemia, irritation, pain, tearing) using ocular tolerability and hyperemia grading scales; and change from baseline for vital signs | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sall Research Medical Center, Artesia, California, United States